CLINICAL TRIAL: NCT03285503
Title: A Single-center, Uncontrolled, Open-label Clinical Trial Evaluating the Pharmacokinetic Characteristics and Safety of Aripiprazole IM Depot in Chinese Patients With Schizophrenia After Multi-dose Administration
Brief Title: PK Study of Aripiprazole IM Depot for Chinese Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 031-403-00049
Record Dates: First submitted 2017-09-11; First posted 2017-09-18 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 400 mg group (Experimental): Aripiprazole IM depot 400mg will be administered every four weeks for 20 weeks after drug switch / steady dose of oral aripiprazole tablets (each subject will receive 5 intramuscular injections totally).
  Interventions: Drug: Aripiprazole IM Depot

INTERVENTIONS:
Drug: Aripiprazole IM Depot — administration of Aripiprazole IM Depot formulation at doses of 400 mg for 5 times in patients with schizophrenia.
  Other Names: ABILIFY MAINTENA

SUMMARY:
This study assess pharmacokinetics and safety of multi-administration of Aripiprazole IM Depot formulation at doses of 400mg in patients with schizophrenia.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics and safety of aripiprazole prolonged IM depot 400mg administered to Chinese adult subjects with schizophrenia every four weeks for 20 consecutive weeks

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, and their legal representatives(or their guardian ), who have signed the informed consent form(ICF);
2. Patients with a diagnosis of schizophrenia as defined by DSM-IV-TR (295.30, 295.10, 295.20,295.90 , 295.60);
3. subjects, both male and female, who are at age between 18 and 64 (also including 18 and 64 years of age) at time of informed consent.

Exclusion Criteria:

1. Presence of other mental disorders than schizophrenia confirmed through diagnostic criteria of DSM-IV-TR;
2. Subjects who are alcoholomania or independent of drug, or have drug abuse history;
3. Positive for any of HIV antibody, HBsAg, HCV antibody and syphilis serology testing;

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to 24 weeks
  To assess the Maximum Plasma Concentration (Cmax) of aripiprazole and its primary metabolite OPC-14857 after administration of the fifth IMD dose.
time of maximum observed plasma concentration (tmax) | up to 24 week
  To assess the time of maximum observed plasma concentration (tmax) of aripiprazole and its primary metabolite OPC-14857 after administration of the fifth IMD dose.
AUC672h | up to 24 weeks
  To assess the time of maximum observed plasma concentration (tmax) of aripiprazole and its primary metabolite OPC-14857 after administration of the fifth IMD dose.
Apparent clearance after extravascular administration | up to 24 weeks
  To assess the apparent clearance after extravascular administration (CL/F) of aripiprazole after administration of the fifth IMD dose.

SECONDARY OUTCOMES:
Adverse Events | up to 24 weeks
  Adverse events will be examined by frequency, severity, seriousness, discontinuation, and relationship to treatment
Vital Signs | up to 24 weeks
  Mean change from baseline and the incidence of potentially clinically relevant abnormal values will be calculated for vital signs
Laboratory Examination | up to 24 weeks
  Mean change from baseline and the incidence of potentially clinically relevant abnormal values will be calculated for routine laboratory tests (including prolactin)

OTHER OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) | up to 24 weeks
  To evaluate the change of Positive and Negative Symptoms Scale (PANSS) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Master, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dong F, Wang F, Yuan X, Zhai Y, Uki M, Jiang T, Li A. Single- and multiple-dose pharmacokinetics, safety, and tolerability of Aripiprazole once-monthly, long-acting intramuscular injection for Chinese adults with schizophrenia. BMC Psychiatry. 2025 Oct 1;25(1):912. doi: 10.1186/s12888-025-07407-w. PMID 41034820